CLINICAL TRIAL: NCT04226144
Title: Comparison Between Breath Stacking Technique Associated With Expiratory Muscle Training and Breath Stacking Technique in Amyotrophic Lateral Sclerosis Patients: a Randomized Single Blind Trial
Brief Title: Breath Stacking Technique Associated With Expiratory Muscle Training in Amyotrophic Lateral Sclerosis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 19 pandemy
Sponsor: Escola Superior de Ciencias da Saude (Other)
Responsible Party: Principal Investigator, Vinicius Zacarias Maldaner da silva, PT, PhD, Escola Superior de Ciencias da Saude
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMTBTALS
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Amyotrophic Lateral Sclerosis; Neuromuscular Diseases
Keywords: respiratory function tests; deglution disorders
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neuromuscular Diseases

STUDY DESIGN:
Intervention Model Description: two-arm, parallel (1:1), superiority, blinded-assessor randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breath Stacking Group (Active Comparator): The lungs are inflated as fully as possible by stacking successive breaths without expiration until the patients' maximal inspiratory capacity (MIC). The participant will be instructed to sustain the air in the lung, closing the glottis. Once the lungs are maximally inflated, the compressed air volume is released under expiratory muscle force, thus generating a cough with lung and chest wall recoil. They will perform 5-8 cycles of breath stacking per session, stacking 3-5 breaths per cycle.
  Interventions: Device: Breath Stacking Group
- Breath stacking and EMT (Experimental): This group will perform the breath stacking technique in addiction with EMT. It will change the one-way valve in this group to VUP (Lumiar, Sao Paulo, Brazil) one-way valve, which allows the patients blow out the air with a counter resistance during all expiratory phase. The initial expiratory pressure will be 8 cmH2O, and could be changed at each visit according to participants' tolerance (either report easy or difficult to exhale assessed by research coordinators. The participants are encouraged to blow out the most slowly that they can do it.
  Interventions: Device: Breath stacking and EMT

INTERVENTIONS:
Device: Breath Stacking Group — Lung recruitment technique using manual bag resuscitation with oronasal mask interface
  Other Names: lung recruitment technique
  Arms: Breath Stacking Group
Device: Breath stacking and EMT — Lung recruitment technique with one way valve with counter resistance during all expiratory phase
  Other Names: VUP
  Arms: Breath stacking and EMT

SUMMARY:
it will be conducted a randomized parallel controlled trial with patients diagnosed with Amyotrophic Lateral Sclerosis (ALS) to compare two techniques to lung recruitment and cough augmentation, to assess their effects on pulmonary function, global functionally, swallowing and ability to speech in these population.

DETAILED DESCRIPTION:
age over 18 years preserved cognition, evidenced by a score greater than or equal to 24 points in the Mini-Mental Status Exam; no barium allergies; without tracheostomy or invasive mechanical ventilation; no diaphragmatic pacemaker and without associated respiratory disease.Participants are excluded if they have pregnancy; previous kidney disease or other concomitant diseases; respiratory diseases and hospitalization in intensive care units (ICUs) during the study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of neuromuscular disease confirmed by neurologists at the referral center for neuromuscular diseases at Brasília prior to screening for recruitment
* age over 18 years
* preserved cognition, evidenced by a score greater than or equal to 24 points in the Mini-Mental Status Exam;
* no barium allergies
* without tracheostomy or invasive mechanical ventilation
* no diaphragmatic pacemaker
* without associated respiratory disease

Exclusion Criteria:

* pregnancy
* previous kidney disease or other concomitant diseases .respiratory diseases and hospitalization in intensive care units (ICUs) during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
maximal respiratory pressures | from baseline to 24 weeks
  change of decline rate of maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) assessed by digital pressure (MVD-500 V.1.1 Microhard System,Porto Alegre, Brazil).
Peak cough flow | from baseline to 24 weeks
  change of decline rate of peak cough flow (PCF) assessed by analogic peak cough flow meter (Respironics-Philips Health Care,PA,USA)
Forced Vital Capacity and Slow Vital Capacity | from baseline to 24 weeks
  Change of decline rate of Forced Vital Capacity (FVC) and Slow Vital Capacity (SVC) predicted by brazilian population assessed by digital spirometer (Vitalgraph, London, UK)

SECONDARY OUTCOMES:
ALSFR-BR | from baseline to 24 weeks
  change of decline rate of Amyotrofic Lateral Sclerosis Functional Revised Scale Brazil (ALSFR-BR)
Voice parameters | from baseline to 24 weeks
  change of Maximum Phonation Time
swalloing function | from baseline to 24 weeks
  change of The Eating Assessment Tool-10 (EAT-10)

CONTACTS AND LOCATIONS:
Overall Officials: Vinicius Maldaner, Principal Investigator — Hospital de Apoio de Brasilia
Locations (1):
- Hospital de Apoio de Brasilia, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dorca A, Alcantara LA, Diniz DS, Sarmet M, Menezes Mateus SR, Franco Oliveira LV, Franco H, Maldaner V. Comparison between breath stacking technique associated with expiratory muscle training and breath stacking technique in amyotrophic lateral sclerosis patients: Protocol for randomized single blind trial. Contemp Clin Trials Commun. 2020 Sep 2;19:100647. doi: 10.1016/j.conctc.2020.100647. eCollection 2020 Sep. PMID 33005816